CLINICAL TRIAL: NCT05862272
Title: A Phase 3B, Single-Arm, Open-Label Study to Evaluate Bone Mineral Density With Long-Term Use of Relugolix Combination Tablet in Premenopausal Women With Heavy Menstrual Bleeding Associated With Uterine Fibroids or Moderate to Severe Pain Associated With Endometriosis
Brief Title: A Phase 3B Study to Evaluate Bone Mineral Density With Long-Term Use of Relugolix Combination Tablet in Women With Uterine Fibroids or Endometriosis
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Sumitomo Pharma Switzerland GmbH (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MVT-601A-006
Record Dates: First submitted 2023-05-08; First posted 2023-05-17 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2025-07

CONDITIONS: Uterine Fibroids; Endometriosis
Keywords: Uterine Leiomyomas; Fibroids; Endometriosis; Bone Mineral Density; Relugolix; Estradiol; Norethindrone acetate
MeSH Terms: conditions — Leiomyoma; Endometriosis; Myofibroma | interventions — relugolix

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Relugolix Combination Tablet (Experimental): Participants will receive relugolix combination therapy orally once daily for 48 months.
  Interventions: Drug: Relugolix Combination Tablet

INTERVENTIONS:
Drug: Relugolix Combination Tablet — A fixed-dose combination tablet containing relugolix 40 mg, estradiol (E2) 1 mg, and norethindrone acetate (NETA) 0.5 mg.
  Other Names: TAK-385; T-1331285; RVT-601; MVT-601; MVT-601A; MYFEMBREE

SUMMARY:
The purpose of this clinical trial to characterize changes in bone mineral density during continuous treatment with relugolix combination tablet for up to 48 months (4 years) and 1 year of post-treatment follow-up in premenopausal women with heavy menstrual bleeding associated with uterine leiomyomas (fibroids) or with moderate-to-severe pain associated with endometriosis.

DETAILED DESCRIPTION:
A prospective, single-arm, open-label, Phase 3B study to assess the effect of continuous 48 months (4 years) of treatment with relugolix combination tablet (relugolix 40 mg/estradiol [E2] 1 mg/norethindrone acetate [NETA] 0.5 mg) on bone mineral density in premenopausal women with heavy menstrual bleeding associated with uterine leiomyomas (fibroids) and premenopausal women with moderate to severe pain associated with endometriosis.

Approximately 1000 women (500 with heavy menstrual bleeding associated with uterine fibroids and 500 with moderate to severe pain associated with endometriosis) will receive relugolix combination tablet, during which time BMD will be assessed by dual-energy X-ray absorptiometry every 6 months.

A subset of participants will be eligible to enter this study following completion of 1 year of treatment with relugolix combination therapy in MVT-601-050 (NCT04756037; SERENE) and will complete 3 years of treatment under this protocol.

Upon completion of 48 months (4 years) of treatment or after early termination of treatment, participants will enter a 1-year post-treatment follow-up period during which time bone mineral density will be assessed at Month 6 and Month 12 following treatment cessation.

ELIGIBILITY:
Key Inclusion Criteria:

* Is a premenopausal woman, 18 to 50 years of age (inclusive);
* A diagnosis of uterine fibroids confirmed by imaging or review of medical records and reports heavy menstrual bleeding negatively affecting quality of life. or
* A diagnosis of endometriosis that is associated with moderate to severe pain.;
* If at risk of pregnancy is willing to avoid pregnancy for 4 years (the duration of the treatment period) using nonhormonal methods of contraception.
* Has a negative serum pregnancy test at the screening visit and a negative urine pregnancy test at the allocation visit (or Month 12 if entering from MVT-601-050 [NCT04756037; SERENE]);
* In good physical and mental health based on medical, surgical, and gynecological history as well as physical, gynecological, and breast examinations, clinical laboratory test results, and vital sign measurements;
* Has a body mass index ≥ 18 kg/m^2.

Key Exclusion Criteria:

* Has a weight or body habitus that exceeds the limit of the DXA scanner or has a condition that precludes an adequate DXA measurement at the lumbar spine or proximal femur
* Has a DXA result demonstrating the following criteria at any anatomic site (lumbar spine, total hip, femoral neck):

  1. For patients entering de novo a Z-score ≤ -1.5 or T-score ≤ -2.0 (if ≥ 40 years of age)
  2. For patients entering from MVT-601-050 (NCT04756037; SERENE) a 12-month on-treatment DXA demonstrating Z-score ≤ -2.0, T-score ≤ -2.5 (if ≥ 40 years of age), or BMD loss ≥ 8% compared with pre-treatment baseline;
* Screening 25-OH vitamin D level < 12 ng/mL (patients with 25-OH vitamin D deficiency with levels ≥ 12 to < 20 ng/mL are permitted if supplementing with vitamin D or if vitamin D supplementation is started in the screening period);
* Has a history of or currently has Cushing's Syndrome, Rheumatoid Arthritis, metabolic bone disease, uncorrected hyperparathyroidism, Paget's disease of the bone, collagen vascular disease, Marfan's syndrome, Ehlers-Danlos syndrome (if confirmed on genetic testing or meets definitive criteria for hypermobility type), chronic kidney disease (CKD) stage 3 or greater with glomerular filtration rate (GFR) < 60 mL/min/m2 using Modification of Diet in Renal Disease (MDRD) method, hyperprolactinemia, known pituitary adenoma, hyperthyroidism, anorexia nervosa, bulimia (within the last year), abnormal bone mineral metabolism (eg, hypophosphatemia). Patients whose hyperparathyroidism or hyperthyroidism has been successfully treated or whose hyperprolactinemia has been successfully treated are allowed;
* History of low trauma (fragility) fracture.
* Past history of use or current use of medication used to treat bone loss other than calcium and vitamin D preparations;
* Prior use of depot-medroxyprogesterone acetate for a treatment period > 2 years (if treatment occurred within the past 5 years) or prior use of GnRH agonist or antagonist for > 12 months total (unless directly entering from MVT-601-050 [NCT04756037; SERENE]);
* Malabsorptive disease (including, but not limited to, inflammatory bowel disease and gastric bypass surgery);
* Current breast cancer, history of breast cancer or other hormone-sensitive malignancy, at increased risk for hormone-sensitive malignancy, or taking an aromatase inhibitor for breast cancer treatment or prevention
* History of organ transplantation or history of bone marrow
* BIRADS ≥ 3 Mammogram at entry (or within the past 6 months).
* Has a known human immunodeficiency virus (HIV) infection or at high risk of contracting HIV
* Has a current psychiatric disorder that would, in the investigator or medical monitor's opinion, impair the ability of the patient to participate in the study or would impair interpretation of their data.
* Is currently using a hormonal intrauterine device or contraceptive implant, hormonal contraceptive, or other prohibited medication and is unwilling to discontinue this hormonal contraception

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 1000 (Estimated)
Dates: Start 2023-08-14 (Actual); Primary Completion 2029-07 (Estimated); Study Completion 2030-09 (Estimated)

PRIMARY OUTCOMES:
Percent change from baseline in BMD (bone mineral density) at Month 48 on-treatment at lumbar spine (L1-L4) in women with uterine fibroids. | Baseline up to Month 48
  Assessed by dual-energy X-ray absorptiometry (DXA) scan.
Percent change from baseline in BMD at Month 48 on-treatment at lumbar spine (L1-L4) in women with endometriosis. | Baseline up to Month 48
  Assessed by dual-energy X-ray absorptiometry (DXA) scan.

SECONDARY OUTCOMES:
Percent change from baseline in BMD at Month 48 on-treatment at total hip and femoral neck in women with uterine fibroids. | Baseline up to Month 48
  Assessed by dual-energy X-ray absorptiometry (DXA) scan.
Percent change from baseline in BMD at Month 48 on-treatment at total hip and femoral neck in women with endometriosis. | Baseline up to Month 48
  Assessed by dual-energy X-ray absorptiometry (DXA) scan.
Percent change from baseline in BMD at Month 6, 12, 18, 24, 30, 36, and 42 on-treatment at the lumbar spine (L1-L4), total hip, and femoral neck in women with uterine fibroids. | Baseline up to Month 6, 12, 18, 24, 30, 36, and 42
  Assessed by dual-energy X-ray absorptiometry (DXA) scan at each designated time points.
Percent change from baseline in BMD at Month 6, 12, 18, 24, 30, 36, and 42 on-treatment at the lumbar spine (L1-L4), total hip, and femoral neck in women with endometriosis. | Baseline up to Month 6, 12, 18, 24, 30, 36, and 42
  Assessed by dual-energy X-ray absorptiometry (DXA) scan at each designated time points.
Percent change from baseline in BMD at Month 48 on-treatment at lumbar spine (L1-L4) in the overall study population. | Baseline up to Month 48
  Assessed by dual-energy X-ray absorptiometry (DXA) scan at each designated time points.
Percent change from baseline in BMD at Month 48 on-treatment at total hip and femoral neck in the overall study population. | Baseline up to Month 48
  Assessed by dual-energy X-ray absorptiometry (DXA) scan at each designated time points.
Percent change from baseline in BMD at Month 6, 12, 18, 24, 30, 36, and 42 on-treatment at the lumbar spine (L1-L4), total hip, and femoral neck in the overall study population. | Baseline up to Month 6, 12, 18, 24, 30, 36, and 42
  Assessed by dual-energy X-ray absorptiometry (DXA) scan at each designated time points.
Percent change from baseline in BMD at post-treatment follow-up (PTFU) Month 6 and PTFU Month 12 at the lumbar spine (L1-L4), total hip, and femoral neck in women with uterine fibroids. | 6 months and 12 months post treatment
  Assessed by dual-energy X-ray absorptiometry (DXA) scan at each designated time points.
Percent change from baseline in BMD at PTFU Month 6 and PTFU Month 12 at the lumbar spine (L1-L4), total hip, and femoral neck in women with endometriosis. | 6 months and 12 months post treatment
  Assessed by dual-energy X-ray absorptiometry (DXA) scan at each designated time points.
Percent change from last on-treatment BMD measurement to PTFU Month 6 and PTFU Month 12 at the lumbar spine (L1-L4), total hip, and femoral neck in women with uterine fibroids. | 6 months and 12 months post treatment
  Assessed by dual-energy X-ray absorptiometry (DXA) scan at each designated time points.
Percent change from last on-treatment BMD measurement to PTFU Month 6 and PTFU Month 12 at the lumbar spine (L1-L4), total hip, and femoral neck in women with endometriosis. | 6 months and 12 months post treatment
  Assessed by dual-energy X-ray absorptiometry (DXA) scan at each designated time points.
Percent change from baseline in BMD at PTFU Month 6 and PTFU Month 12 at the lumbar spine (L1-L4), total hip, and femoral neck in the overall study population. | 6 months and 12 months post treatment
  Assessed by dual-energy X-ray absorptiometry (DXA) scan at each designated time points.
Percent change from last on-treatment BMD measurement to PTFU Month 6 and PTFU Month 12 at the lumbar spine (L1-L4), total hip, and femoral neck in the overall study population. | 6 months and 12 months post treatment
  Assessed by dual-energy X-ray absorptiometry (DXA) scan at each designated time points.
Incidence of treatment-emergent serious adverse events, and non-serious adverse events leading to treatment discontinuation or withdrawal from the study during the 48 months of treatment. | Baseline up to Month 48
  Safety analyses will be conducted by each safety population: 1) women with uterine fibroids, 2) women with endometriosis, and 3) overall population. The treatment-emergent period will be defined as the period of time from the date of the first dose of the study drug through 14 days after the last dose of study drug, or the date of initiation of another investigational agent or hormonal therapy affecting the hypothalamic-pituitary gonadal axis or surgical intervention for uterine fibroids or for endometriosis, whichever occurs first.
Incidence and location of fractures during the 48 months on treatment and 12 months PTFU. | Baseline up to Month 48 and 12 months post treatment
  Safety analyses will be conducted by each safety population: 1) women with uterine fibroids, 2) women with endometriosis, and 3) overall population. All adverse events will be coded to preferred term and system organ class using Medical Dictionary for Regulatory Activities (MedDRA) version 24.0 or higher. The incidence of fractures will also be summarized by anatomical sites and whether the fracture qualifies as a fragility fracture. A participant reporting the same adverse event more than once is counted once, and at the maximum severity or strongest relationship to study drug treatment when calculating incidence.

CONTACTS AND LOCATIONS:
Overall Officials: Myovant Medical Director, Study Director — Myovant Sciences GmbH
Locations (102):
- United States (102):
  - Mobile, Mobile, Alabama
  - Chandler, Chandler, Arizona
  - Mesa, Mesa, Arizona
  - Peoria, Peoria, Arizona
  - Phoenix, Phoenix, Arizona
  - Tucson, Tucson, Arizona
  - Burbank, Burbank, California
  - Canoga Park, Canoga Park, California
  - Encinitas, Encinitas, California
  - Inglewood, Inglewood, California
  - Lomita, Lomita, California
  - Long Beach, Long Beach, California
  - Los Angeles, Los Angeles, California
  - Sacramento, Sacramento, California
  - San Fernando, San Fernando, California
  - Stanford, Stanford, California
  - Valley Village, Valley Village, California
  - Aurora, Aurora, Colorado
  - Greenwood Village, Greenwood Village, Colorado
  - Lakewood, Lakewood, Colorado
  - Washington, Washington D.C., District of Columbia
  - Aventura, Aventura, Florida
  - Deland, DeLand, Florida
  - Hialeah, Hialeah, Florida
  - Kissimmee, Kissimmee, Florida
  - Lake Worth, Lake Worth, Florida
  - Margate, Margate, Florida
  - Miami, Miami, Florida
  - Miami Beach, Miami Beach, Florida
  - Miami Springs, Miami Springs, Florida
  - New Port Richey, New Port Richey, Florida
  - Orlando, Orlando, Florida
  - Panama City, Panama City, Florida
  - Sarasota, Sarasota, Florida
  - Tamarac, Tamarac, Florida
  - Tampa, Tampa, Florida
  - Venice, Venice, Florida
  - West Palm Beach, West Palm Beach, Florida
  - Atlanta, Atlanta, Georgia
  - College Park, College Park, Georgia
  - Fayetteville, Fayetteville, Georgia
  - Norcross, Norcross, Georgia
  - Idaho Falls, Idaho Falls, Idaho
  - Meridian, Meridian, Idaho
  - Chicago, Chicago, Illinois
  - Schaumburg, Schaumburg, Illinois
  - Lenexa, Lenexa, Kansas
  - Wichita, Wichita, Kansas
  - Covington, Covington, Louisiana
  - Marrero, Marrero, Louisiana
  - Metairie, Metairie, Louisiana
  - New Orleans, New Orleans, Louisiana
  - Slidell, Slidell, Louisiana
  - Baltimore, Baltimore, Maryland
  - Laurel, Laurel, Maryland
  - Towson, Towson, Maryland
  - Bay City, Bay City, Michigan
  - Dearborn Heights, Dearborn Heights, Michigan
  - Detroit, Detroit, Michigan
  - Ridgeland, Ridgeland, Mississippi
  - Saint Louis, St Louis, Missouri
  - St Louis, St Louis, Missouri
  - Grand Island, Grand Island, Nebraska
  - Norfolk, Norfolk, Nebraska
  - Las Vegas, Las Vegas, Nevada
  - North Las Vegas, North Las Vegas, Nevada
  - West New York, West New York, New Jersey
  - Durham, Durham, North Carolina
  - New Bern, New Bern, North Carolina
  - Raleigh, Raleigh, North Carolina
  - Winston Salem, Winston-Salem, North Carolina
  - Cincinnati, Cincinnati, Ohio
  - Cleveland, Cleveland, Ohio
  - Columbus, Columbus, Ohio
  - Dublin, Dublin, Ohio
  - Englewood, Englewood, Ohio
  - Middletown, Middletown, Ohio
  - Erie, Erie, Pennsylvania
  - Philadelphia, Philadelphia, Pennsylvania
  - Bluffton, Bluffton, South Carolina
  - Greenville, Greenville, South Carolina
  - Summerville, Summerville, South Carolina
  - West Columbia, West Columbia, South Carolina
  - Chattanooga, Chattanooga, Tennessee
  - Jackson, Jackson, Tennessee
  - Memphis, Memphis, Tennessee
  - Arlington, Arlington, Texas
  - Dallas, Dallas, Texas
  - Fort Worth, Fort Worth, Texas
  - Galveston, Galveston, Texas
  - Houston, Houston, Texas
  - League City, League City, Texas
  - Pearland, Pearland, Texas
  - San Antonio, San Antonio, Texas
  - Sugar Land, Sugar Land, Texas
  - Webster, Webster, Texas
  - Pleasant Grove, Pleasant Grove, Utah
  - Salt Lake City, Salt Lake City, Utah
  - Annandale, Annandale, Virginia
  - Newport News, Newport News, Virginia
  - Virginia Beach, Virginia Beach, Virginia
  - Seattle, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No